CLINICAL TRIAL: NCT04862650
Title: A Phase II Trial of the Efficacy and Safety of the Combination of Cemiplimab and Low-Dose Paclitaxel and Carboplatin in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cemiplimab, Low-Dose Paclitaxel and Carboplatin for the Treatment of Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marcelo Bonomi (Other)
Responsible Party: Sponsor-Investigator, Marcelo Bonomi, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-20258; NCI-2021-02081 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-03-26; First posted 2021-04-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Oral Cavity Squamous Cell Carcinoma; Metastatic Oropharyngeal Squamous Cell Carcinoma; Pathologic Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Unknown Primary; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8; Stage IVC Hypopharyngeal Carcinoma AJCC v8; Stage IVC Laryngeal Cancer AJCC v8; Stage IVC Lip and Oral Cavity Cancer AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms | interventions — Carboplatin; cemiplimab; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cemiplimab, paclitaxel, carboplatin) (Experimental): Patients will be treated with a combination of cemiplimab 350 mg every three weeks, with weekly combination of paclitaxel 25 mg/m2 and carboplatin AUC 1. Treatment will continue for a total of 24 months or until disease progression or unacceptable toxicity. Weekly chemotherapy will stop after six months of treatment (24 weeks). A ten patient safety run-in phase will be initially performed.
  Interventions: Drug: Carboplatin; Biological: Cemiplimab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN2810
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II trial studies the effect of cemiplimab in combination with low-dose paclitaxel and carboplatin in treating patients with squamous cell carcinoma of the head and neck that has come back (recurrent) or spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as cemiplimab , may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, like paclitaxel and carboplatin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving cemiplimab in combination with paclitaxel and carboplatin may work better in treating recurrent or metastatic squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the overall response rate (ORR) at 12 weeks of treatment with the treatment combination cemiplimab, paclitaxel, and carboplatin.

SECONDARY OBJECTIVES:

I. To assess toxicity/tolerance to the proposed treatment combination (a safety run-in phase of ten patients will be performed initially).

II. To assess progression-free survival (PFS) and overall survival (OS) at one and two years.

EXPLORATORY OBJECTIVES:

I. Prospectively test the ability of our clinical nomogram to predict median OS in squamous cell carcinoma of the head and neck (SCCHN) patients planning to receive first-line cemiplimab in combination with low-dose weekly paclitaxel and carboplatin.

II. To assess the PFS and OS of patients with combined positive score (CPS) <1%, >1%, and > 20%.

III. Compare the predictive power of our nomogram to that of CPS in the prospective cohort, as well as evaluate the combined correlation of nomogram and CPS to median OS.

IV. Perform comprehensive immune analysis including phenotypic analysis of immune cell subsets using high dimensional spectral flow cytometry. T cell functionality and ability to produce cytokines after ex vivo stimulation for all T cells and E6/E7-reactive T cells (P16+ subset patients) and TCR sequencing to determine if clonal T cell populations emerge from the tumor of responding patients in comparison with non-responders.

OUTLINE:

Patients receive cemiplimab intravenously (IV) over 30 minutes every 3 weeks (Q3W) for up to 104 weeks, and paclitaxel IV over 60 minutes and carboplatin IV over 30 minutes once weekly (QW) for up to 24 weeks. Treatment continuous in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 14 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent/metastatic (R/M) SCCHN of the oral cavity, oropharynx, larynx and hypopharynx
* No prior systemic therapy for treatment of R/M disease
* Patients with squamous cell carcinoma of an unknown primary are eligible provided their tumor tested positive for p-16 and they have previously received treatment for locoregional head and neck cancer
* Must be at least four weeks since prior radiation and/or surgery
* Must be at least four weeks from curative intent systemic therapy. Of note: patients who have received up to two courses of chemoradiotherapy (CRT) for locoregionally advanced disease are eligible. Induction chemotherapy will not be considered a separate line of therapy
* At least one measurable lesion as defined by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 on screening computed tomography (CT) or magnetic resonance imaging (MRI)
* 18 years of age and older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* White blood cell (WBC) count > 2,500 cells/uL
* Absolute neutrophil count (ANC) >1,500 cells/uL
* Platelet count >= 100,000 cells/uL
* Hemoglobin >= 9 g/dL
* Creatinine =< 1.6 mg/dL
* Total bilirubin =< 1.6 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate transaminase [AST]), serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x upper limit of normal (ULN)
* Potassium >= lower limit of normal (LLN)
* Willingness to use medically acceptable contraception throughout the study period and four months after the final administration of treatment
* For female subjects with reproductive potential: a negative serum pregnancy test at baseline
* Ability and willingness to provide written informed consent and to comply with the study visits and assessment schedule

Exclusion Criteria:

* Disease amenable to curative local therapy
* Nasopharyngeal, salivary gland, lip, or sinonasal carcinoma
* Disease that requires corticosteroids or other ongoing immunosuppressive treatment
* Previous treatment with mAb-based immunotherapy for treatment of prior oncologic treatment
* Previous treatment with PI3K inhibitors
* Known brain metastases, unless stable for at least 21 days prior to registration
* Known infection human immunodeficiency virus (HIV), hepatitis B or C
* Clinically significant cardiac disease (e.g., congestive heart failure, unstable or uncontrolled angina, myocardial infarction) within the past six months
* History of pneumonitis within the past five years
* Recipient of live vaccines (including attenuated) within 30 days of planned study treatment
* Female patients who are pregnant or breast-feeding
* Any other condition or circumstance that could interfere with adherence to the study's procedures or requirements or otherwise compromise the study's objectives in the opinion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 12 weeks
  ORR defined as the proportion of patients with a documented complete response (CR) + partial response (PR) at week 12 of treatment based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. An ORR of 40% (percent) or higher will be consider a positive result. Simon two-stage optimal design will be used.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of enrollment until documented disease progression, assessed up to 2 years
  PFS will be calculated based on RECIST criteria.
Overall survival (OS) | From the date of patient enrollment into the trial until death, assessed up to 2 years
Incidence of adverse events | Up to 24 weeks
  Toxicity will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
Ability of our clinical nomogram to predict median OS in squamous cell carcinoma of the head and neck patients planning to receive first-line cemiplimab in combination with low-dose weekly paclitaxel and carboplatin | Up to 24 weeks
PFS of patients with combined positive score (CPS) < 1%, > 1%, and > 20% | Up to 2 years
OS of patients with CPS < 1%, > 1%, and > 20% | Up to 2 years
Predictive power of our nomogram to that of CPS in the prospective cohort, as well as evaluate the combined correlation of nomogram and CPS to median OS | Up to 24 weeks
Comprehensive immune analysis | Up to 24 weeks
  The analysis of T cell receptor (TCR) repertoires will be performed using R package 'divo.' The diversity of TCR repertoires will be assessed using Renyi entropy. Longitudinal changes of TCR repertoire will be analyzed using Morisita-Horn Index by comparing the similarity (distance) between the repertoire in each time point and the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo R Bonomi, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu